CLINICAL TRIAL: NCT05832567
Title: Mechanisms of Open and Hidden Placebo in Stroke Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director of Spaulding Neuromodulation Center, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2023P000884
Record Dates: First submitted 2023-03-24; First posted 2023-04-27 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke; placebo
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Active rTMS (Active Comparator): The participant will receive a session of low frequency rTMS to the contralesional primary motor cortex. Low frequency rTMS stimulation will be applied according to the following parameter: intensity of 80% MT (intensity could be adjusted if not comfortable to the subject), frequency of 1 Hz, 1200 pulses as a single, continuous train lasting 20 minutes.
  Interventions: Device: Active rTMS
- Sham rTMS (Sham Comparator): The investigators will place the coil in the same location, usually used for the active stimulation with the same stimulation parameters. However, the investigators will replace the active coil with a sham coil to ensure no stimulation is provided.
  Interventions: Device: Sham rTMS
- Open Placebo (Placebo Comparator): The open placebo will consist of typical prescription medicine bottle of placebo pills with a label clearly marked "placebo pills" "take 2 pills twice daily." The placebo pills are made from Microcrystalline Cellulose.
  Interventions: Dietary Supplement: Open Placebo
- No Intervention (No Intervention): It consists of treatment-as-usual group.

INTERVENTIONS:
Device: Active rTMS — Subjects will undergo repetitive transcranial magnetic stimulation, each session lasting 20 minutes.
  Arms: Active rTMS
Device: Sham rTMS — Subjects will undergo sham repetitive transcranial magnetic stimulation, each session lasting 20 minutes.
  Arms: Sham rTMS
Dietary Supplement: Open Placebo — The open placebo will consist of an inactive substance pill commonly used in clinical trials and given to the subject in a regular pill dispenser.
  Arms: Open Placebo

SUMMARY:
This trial aims to investigate whether placebo in isolation (open and hidden) has a specific neural signature in stroke subjects thus providing a novel mechanism to explain placebo effects that can be used to ultimately enhance stroke rehabilitation therapies.

DETAILED DESCRIPTION:
Placebo effect leads to significant effects on brain excitability and connectivity, ultimately influencing clinical outcomes, including motor learning in stroke. This trial will provide critical mechanistic data to improve the understanding of placebo in stroke clinical trials, as to solve methodological and ethical dilemma in research designs, and to improve its clinical outcomes. It aims to investigate whether placebo in isolation (open and hidden) has a specific neural signature in stroke subjects. For this purpose, the investigators plan to recruit 56 chronic stroke participants, that will be randomized using blocked randomization in a 2:2:2:1 proportion to one of the following groups, respectively: 1) open placebo (OP) alone (16 subjects); 2) sham rTMS alone (16 subjects); 3) no intervention (16 subjects); or 4) active rTMS alone (8 subjects). All four groups will undergo 2 weeks of daily intervention visits (10 sessions).

ELIGIBILITY:
Inclusion Criteria:

1. Adults with hemiparesis due to chronic stroke
2. Stroke duration of 6 months or more
3. Fugl-Meyer scale upper extremity motor assessment score of > 11 and ≤ 56
4. Pre-stroke disability (defined as a score of < 3 on the Modified Rankin Scale)
5. Age 18 or older

Exclusion Criteria:

1. Stroke of anterior cerebral artery territory with prefrontal lesion and stroke-related decreased EEG power in the prefrontal cortex
2. Unable to understand instructions
3. TMS contraindications: electronic hardware in close contact to the discharging coil such as cochlear implant, internal pulse generator or medical pump
4. Concurrent unstable medical conditions
5. A score of 24 or higher on the Hamilton Depression Rating Scale (HDRS)
6. Joint or paretic extremity pain likely to interfere with assessments
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG): Frontal alpha asymmetry | Change from 2 weeks to baseline
  The FAA score will be calculated by subtracting the natural log-transformed alpha power in the left frontal region (F3, F7, Fp1) from the natural log-transformed power in the right frontal region (F4, F8, Fp2).

SECONDARY OUTCOMES:
Fugl-Meyer motor scale (FM) | Change from 2 weeks to baseline
  The investigators will use this tool for motor function after stroke. It is valid, responsive to change, and widely used for motor function and recovery assessment in stroke patients. Items are scored on a 3-point ordinal scale, being 0 the lowest and 2 the highest value. A higher score means a better outcome.
Premotor-M1 (PM-M1) connectivity | Change from 2 weeks to baseline
  For the PM-M1 connectivity computation, the investigators will calculate the spectral coherence score, which indicates the functional connectivity in brain activity between two cortical regions and is calculated as a function of frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital/Harvard Medical School
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No